CLINICAL TRIAL: NCT07254533
Title: Diagnosis and Quantification of Hepatic Steatosis Using Near-infrared Spectroscopy
Acronym: STEATO-NIR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RCAPHM24_0352; 2024-A02004-43 (Other: IDRCB)
Record Dates: First submitted 2025-11-17; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Hepatic Transplantation; Steatohepatitis
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- liver grafts (Experimental)
  Interventions: Device: Near-infrared spectrometer
- Surgical specimens (hepatectomy) (Experimental)
  Interventions: Device: Near-infrared spectrometer

INTERVENTIONS:
Device: Near-infrared spectrometer — Scan of the liver via near-infrared spectrometer

SUMMARY:
In liver transplantation, the main problem is the shortage of grafts due to the small pool of donors. In order to increase the number of donors, grafts are increasingly being taken from older donors, known as 'expanded criteria' donors, who have liver steatosis lesions. Currently, expanded criteria donors account for 75% of liver transplants, whereas in 2009 they accounted for less than 30% of liver transplants.

Steatosis and its progression Non-alcoholic steatohepatitis (NASH) is an emerging disease in industrialised countries due to obesity, and corresponds to the accumulation of intracytoplasmic triglycerides.

Steatosis is diagnosed when this fat content represents more than 5% of the total liver mass. There are two types of steatosis: microvesicular steatosis and macrovacuolar steatosis, defined by the presence of lipid droplets larger than the nucleus with a nucleus displaced to the periphery. Macrovacuolar steatosis is responsible for impaired liver function if it is present in ≥30% of hepatocytes. It is a factor in poor prognosis for liver transplants, with reduced graft and recipient survival and an increase in early graft dysfunction after liver transplantation. The quantification of hepatic steatosis is based on the pathological analysis of a liver biopsy, which is currently the gold standard.

This technique has disadvantages: it is an invasive method, requiring an experienced pathologist, and presents inter-individual variability in the assessment and quantification of steatosis.

It is therefore essential to develop new non-invasive diagnostic tools that can identify the presence of steatosis > 5% and ≥ 30%. Several non-invasive techniques for diagnosing steatosis have been studied: Fibroscan, CT scan, MRI, but none of those studied previously allow for the accurate quantification of hepatic steatosis, particularly macrovacuolar steatosis, with instant results.

ELIGIBILITY:
Inclusion Criteria:

Liver grafts:

* Men or women aged 18 and over
* All donors accepted by the MA4FC procurement team, including brain-dead donors and Maastricht 3 donors, even if placed on a perfusion machine
* Donors whose families have received information about the study and have not expressed any opposition

Surgical specimens (hepatectomy):

* Men or women aged 18 years and older
* Subjects who have undergone surgery for any indication of hepatectomy
* Affiliated with social security,
* Having received information about the study and not having expressed opposition

Exclusion Criteria:

Liver grafts:

* Donors whose liver will be subject to a SPLIT procedure
* Donors for whom there is a medical-legal obstacle
* Donors whose family or loved ones oppose scientific sampling: The hospital coordination team will consult the national refusal register and question loved ones to determine whether the deceased would have opposed sampling. If the donor and/or family oppose scientific sampling, then sampling will not be performed.

Surgical specimens (hepatectomy):

* Subjects covered by Articles L1121-5 to 1121-8 of the Public Health Code (minors, adults under guardianship or curatorship, patients deprived of their liberty, pregnant or breastfeeding women),
* Subjects who do not understand the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Sensibility of near-infrared spectroscopy | through study completion, an average of 1 year
  Estimate the performance of near-infrared spectroscopy for quantifying hepatic steatosis (>5%).

SECONDARY OUTCOMES:
Specificity of the near-infrared spectroscopy | From enrollement to the end of the study at 12 months
Youden's index of the near-infrared spectroscopy | From enrollement to the end of the study at 12 months
Likelihood index + and - of the near-infrared spectroscopy | From enrollment to the end of the study at 12 months
Nanogram likelihood ratio of the near-infrared spectroscopy | From enrollement to the end of the study at 12 months
ROC curve of the near-infrared spectroscopy | From enrollement to the end of the study at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Timone Hospital, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided